CLINICAL TRIAL: NCT00686283
Title: Personalized Exercise for Adolescents With Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Melissa Faulkner, Associate Dean, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RNR009267B; 7R21NR009267-02 (NIH)
Record Dates: First submitted 2008-05-20; First posted 2008-05-29 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes
Keywords: Adolescents; Diabetes; Exercise
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise prescription (Other): Each adolescents with type 1 or type 2 diabetes received individual fitness testing and a personalized exercise program prescription developed by an exercise physiologist. Pretest and posttest measures of glucose control and cardiorespiratory fitness, heart rate variability, metabolic control, lipid profile, body composition, and inflammatory markers, as well as psychological outcomes (i.e., diabetes quality of life) were completed.
  Interventions: Behavioral: PEP intervention

INTERVENTIONS:
Behavioral: PEP intervention — This study will explore the feasibility of adherence to a personalized exercise prescription (PEP) in adolescents with type 1 or type 2 diabetes. The PEP intervention consists of a 2-hour group education session and a 16-week personalized exercise plan implemented in the home or community setting with the use of parental support and care ambassadors. Care ambassadors will maintain consistency of interactions with specific families for the duration of the PEP intervention. This consistency will aid in establishing rapport with the adolescents and parents to answer any questions and provide guidance for adhering to the PEP plan. The PEP intervention will be mutually planned with each teen and parent based upon the assessment of the teen's personal and cultural choices, including family and community resources. Exercise frequency, duration, and intensity for the teen with diabetes will be documented with a MTI ActiGraph accelerometer (Fort Walton Beach, FL).

SUMMARY:
This study aims to determine the likely benefits of a study that would use the novel techniques both of writing an exercise "prescription" and of including the family and/or community in sticking to the exercise prescription by youths with diabetes, who often suffer eventual cardiovascular complications that might be lessened by the exercise.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is now the sixth leading cause of death in the U.S., primarily due to cardiovascular (CV) complications. People with DM have a 2 to 4 times increased risk for heart disease. An increasing number of adolescents are diagnosed with DM, predisposing them to CV morbidity and mortality in early adulthood. Using a comparison group pretest-posttest design, the Primary Aim of this investigation is to determine the feasibility of conducting a novel personalized exercise prescription (PEP) intervention with 20 adolescents who have type 1 DM and 20 adolescents with type 2 DM. We will explore the influence of DM-specific family social support, exercise self-efficacy, and benefits and barriers to exercise on adherence to PEP. The Secondary Aim is to explore possible changes in physiological (i.e., cardiorespiratory fitness, heart rate variability, metabolic control, and lipid profile) and psychological outcomes (i.e., diabetes quality of life [QOL]) of the PEP intervention in adolescents with type 1 or type 2 DM. Long-term benefits of exercise for persons with DM include decreased risk factors for CV disease, improved well-being, and increased life expectancy. The current decline in physical activity during adolescence is problematic, particularly for those with DM, who have an added risk for future CV disease. The limited research available on the efficacy of exercise interventions with youths who have type 1 DM indicates improvements in cardiorespiratory fitness, lipid profile, and glucose regulation. No published exercise intervention research with adolescents who have type 2 DM is available. However, exercise interventions with overweight youth have shown increased heart rate variability and cardiorespiratory fitness. Although numerous studies have examined various school-based strategies to promote more physically active lives in youth populations, no studies have examined the feasibility of conducting individualized, culturally focused exercise prescriptions for adolescents with type 1 or type 2 DM that incorporate family support in a home or community setting. Nor have studies addressed the possible psychosocial and physiological outcomes of these personalized approaches. This investigation will extend the principal investigator's program of research that identified differences in CV risks for adolescents with type 1 vs. type 2 DM. Determining factors that influence the conduct and outcomes of individualized exercise interventions for adolescents with DM can potentially lead to the development of programs that promote adherence to exercise, avert complications, and improve QOL and overall health.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12 to 19
* With a diagnosis of type 1 or type 2 DM
* Score on Physical Activity Recall (PAR) Scale of 36 metabolic equivalents (METs) or less to ensure enrollment of youths who are not already engaged in a regular exercise or sports program
* Have a parent (guardian) who also agrees to attend personalized exercise program (PEP) training, participate in exercising and provide ongoing encouragement and support for PEP, and who does not have any positive responses to the Physical Activity Readiness Questionnaire (PAR-Q). The decision to use a value for METs < 36 is based upon current PAR data from the PI's R01 that revealed a mean score of 34.7 ± 3.1 for teens with type 1 DM and 33.5 ± 1.4 for teens with type 2 DM. Mean scores for both groups reflect activity levels that are well below the current recommendation of 60 minutes of moderate to vigorous exercise on most days of the week.

Exclusion criteria:

Subjects will be excluded if they:

* Are in a school grade that is not appropriate to age within 2 years (this is to control for overt delays in cognition, literacy, and psychological or behavioral functioning)
* Have developed diabetes as a secondary condition to treatment for another chronic condition (i.e., cancer)
* Have known cardiac defects
* Are pregnant females.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2007-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
exercise adherence | Longitudinal and following the 16-week intervention

SECONDARY OUTCOMES:
cardiorespiratory fitness | Following the 16-week intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center, Tucson, Arizona, United States

REFERENCES:
- [Derived] Michaliszyn SF, Higgins M, Faulkner MS. Patterns of Physical Activity Adherence by Adolescents With Diabetes or Obesity Enrolled in a Personalized Community-Based Intervention. Diabetes Educ. 2018 Dec;44(6):519-530. doi: 10.1177/0145721718805693. Epub 2018 Oct 11. PMID 30306834
- [Derived] Faulkner MS, Michaliszyn SF, Hepworth JT, Wheeler MD. Personalized exercise for adolescents with diabetes or obesity. Biol Res Nurs. 2014 Jan;16(1):46-54. doi: 10.1177/1099800413500064. Epub 2013 Aug 20. PMID 23965300
- [Derived] Michaliszyn SF, Faulkner MS. Physical activity and sedentary behavior in adolescents with type 1 diabetes. Res Nurs Health. 2010 Oct;33(5):441-9. doi: 10.1002/nur.20393. PMID 20672318